CLINICAL TRIAL: NCT02917616
Title: The Effect of Drinking-Water pH on the Human Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-15011825
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alkaline water (Experimental): Two liters (minimum) daily of alkaline drinking-water (pH=9) for 14 days
  Interventions: Other: Alkaline drinking-water
- Neutral Water (Active Comparator): Two liters (minimum) daily of neutral drinking-water (pH=7) for 14 days
  Interventions: Other: Neutral drinking-water

INTERVENTIONS:
Other: Alkaline drinking-water
  Arms: Alkaline water
Other: Neutral drinking-water
  Arms: Neutral Water

SUMMARY:
This study evaluates the effect of alkaline (pH=9) versus neutral (pH=9) drinking-water on the gut microbiota of healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Non-smoker
* Age 18 - 35 years
* Weight stabile for at least 2 months
* BMI between 20.0 - 27.0 kg/m^2

Exclusion Criteria:

* Habitual consumption of caloric or artificially sweetened beverages in excess of 1L/week
* Habitual average consumption of alcohol in excess of 7 drinks/week
* Antibiotic treatment within two months of inclusion
* Chronic or acute illness
* Previous abdominal surgery

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Shannon's alpha diversity index | Intervention day 14
  Diversity of the gut microbial community

SECONDARY OUTCOMES:
Simpsons' reciprocal diversity index | Intervention day 14
  Diversity of the gut microbial community
Observed richness | Intervention day 14
  Observed number of operational taxonomic units
Estimated richness | Intervention day 14
  Number of operational taxonomic units estimated using the Chao1 method
Unweighted UniFrac | Intervention day 14
  Inter-individual diversity of the gut microbial community assessed using principal coordinate ordination of unweighted UniFrac distances
Weighted UniFrac | Intervention day 14
  Inter-individual diversity of the gut microbial community assessed using principal coordinate ordination of weighted UniFrac distances
Bray-Curtis | Intervention day 14
  Inter-individual diversity of the gut microbial community assessed using principal coordinate ordination of Bray-Curtis distances
Operational taxonomic unit | Intervention day 14
  Relative abundance of individual operational taxonomic units
Bacterial genera | Intervention day 14
  Relative abundance of operational taxonomic units aggregated at genus level
Plasma glucose; global | Intervention day 14
  Global test of intervention effect on plasma glucose concentration during an oral glucose tolerance test
Serum insulin; global | Intervention day 14
  Global test of intervention effect on serum insulin concentration during an oral glucose tolerance test
Serum insulin; individual timepoints | Intervention day 14
  Intervention effect on serum insulin concentration at individual timepoints druing an oral glucose tolerance test
Plasma glucose; individual timepoints | Intervention day 14
  Intervention effect on plasma glucose concentration at individual timepoints druing an oral glucose tolerance test
High sensitivity C-reactive protein | Intervention day 14

CONTACTS AND LOCATIONS:
Overall Officials: Oluf Pedersen, MD, DMSc, Principal Investigator — The Novo Nordisk Foundation Center for Basic Metabolic Research

IPD SHARING:
Plan to Share IPD: Yes
Anonymised datasets generated during the current study are available from the corresponding author on reasonable request

REFERENCES:
- [Derived] Hansen TH, Thomassen MT, Madsen ML, Kern T, Bak EG, Kashani A, Allin KH, Hansen T, Pedersen O. The effect of drinking water pH on the human gut microbiota and glucose regulation: results of a randomized controlled cross-over intervention. Sci Rep. 2018 Nov 9;8(1):16626. doi: 10.1038/s41598-018-34761-5. PMID 30413727